CLINICAL TRIAL: NCT05233722
Title: Mechanistic Target of Rapamycin (mTOR) as Mediator of Exercise-induced Insulin Sensitivity Study
Brief Title: mTOR as Mediator of Insulin Sensitivity Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Danish Diabetes Academy (Other)
Responsible Party: Principal Investigator, Professor Jorgen FP Wojtaszewski, Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Rapa Study
Record Dates: First submitted 2022-01-17; First posted 2022-02-10 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Insulin Sensitivity
Keywords: Exercise; Muscle insulin Sensitivity; Muscle Glucose uptake; Muscle protein synthesis; mTOR
MeSH Terms: conditions — Insulin Resistance; Motor Activity | interventions — Exercise; Insulin Infusion Systems; Sirolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The participant will be blinded upon receiving the drug. 4-5 researchers will conduct various measurements on the subject upon each experimental day. Only the clinical responsible will know which drug is administered, while the remaining researchers will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-exercise insulin sensitivity following placebo administration (Placebo Comparator): Young healthy males will ingest placebo (blinded) and perform a single bout of knee-extensor exercise and insulin action is investigated 4 hours after cessation of exercise. Insulin action towards muscle glucose uptake and protein synthesis will be investigated during a 120 min euglycemic hyperinsulinemic clamp.
  Interventions: Other: Exercise; Procedure: Insulin infusion; Drug: Placebo
- Post-exercise insulin sensitivity following Rapamycin administration (Experimental): Young healthy males will ingest Rapamycin (blinded) and perform a single bout of knee-extensor exercise and insulin action is investigated 4 hours after cessation of exercise. Insulin action towards muscle glucose uptake and protein synthesis will be investigated during a 120 min euglycemic hyperinsulinemic clamp.
  Interventions: Other: Exercise; Procedure: Insulin infusion; Drug: Rapamycin

INTERVENTIONS:
Other: Exercise — 1 hour of one-legged knee-extensor exercise followed by 4 hours of rest
Procedure: Insulin infusion — 2 hours of Euglycemic Hyperinsulinemic Clamp
Drug: Placebo — Administration of 800 mg of calcium tablets
  Arms: Post-exercise insulin sensitivity following placebo administration
Drug: Rapamycin — Administration of 16 mg of Rapamycin tablets
  Arms: Post-exercise insulin sensitivity following Rapamycin administration

SUMMARY:
The study investigates the role of mTOR in mediating enhancement of muscle insulin sensitivity following a single bout of exercise.

This will be investigated in young healthy male subjects by administering the pharmacological mTOR inhibitor Rapamycin in a crossover blinded experimental setup known to enhance muscle insulin sensitivity following one-legged knee-extensor exercise.

DETAILED DESCRIPTION:
Trial A: During trial A the study subject will arrive at the research laboratory and eat a morning meal at 6:30 a.m. corresponding to 5% of the daily energy requirements. It is requested that the study subject will arrive in a car or with public transportation. At the same time, the subject will ingest 16 mg of Rapamycin or placebo (800 mg Calcium) in pill form. Following ingestion, the study subject will rest for 2 hour and at that time catheters are inserted in both femoral veins, the femoral artery in one of the legs and in each forearm vein (antecubital veins) for later blood sampling and intravenous infusion of insulin, glucose, stable D2-glucose and stable 13C6-phenylalanine. At 8:30 a.m. the study subjects will perform one-leg knee extension exercise for 1 hour at an intensity of 80% of maximal work capacity. In this work protocol there are inserted 3 intervals of 5 minutes duration where the study subject works at 100% of maximal intensity with the purpose of securing a full activation/recruiting of all muscle fibers. Immediately following conclusion of the exercise bout 13C6-phenylalanine is infused for later determination of muscle protein synthesis. 2 hours into the recovery from exercise D2-glucose is infused for later determination of hepatic glucose production. 4 hours into the recovery from exercise an euglycaemic hyperinsulinemic clamp will be initiated for 2 hours for determination of insulin stimulated muscle glucose uptake. Muscle biopsies from the m. vastus lateralis muscle in one or both legs will be taken before, immediately after, as well as 2, 4 and 6 hours after conclusion of exercise. Pulmonary oxygen uptake is measured with the use of an online system before, during and after exercise and is used for determination of substrate metabolism. Blood samples from the femoral veins in both legs and the femoral artery in one of the legs are drawn before, during exercise, and during the recovery period after exercise. At the same time blood flow is measured in the femoral arteries in both legs with the use of Doppler technique. Determination of arteriovenous difference (AV difference) by simultaneous measurement of blood flow enables us to calculate skeletal muscle glucose uptake and uptake/release of relevant substances (proteins, peptides and metabolites etc.). The experimental part of trial A is completed at 15:30 p.m. The study subject will be given food and drink and will be observed for one hour before they may leave the research laboratory.

Trial B is an identical protocol, except that the subject will receive opposite drug from trial A (Rapamycin or placebo). Trial A and B will be separated by a minimum of 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons (no known disease) without diabetes in the family
* No use of medications
* Non-smokers
* Men
* Age 22-35 years
* Physical activity level (VO2peak) between 30-50 mL O2/min/kg
* BMI between 18.0 and 25.0

Exclusion Criteria:

* Women
* Physical activity (e.g., running, cycling, fitness, etc.) above 6 hours a week.
* Persons who show signs of metabolic diseases, hematologic diseases, reduced liver function, human immunodeficiency virus (HIV), hepatitis, thyroid diseases or other signs of disease that may affect the outcome of the study or the study subject's wellbeing will be excluded.
* Acute sickness less than 2 weeks prior to study start.
* If disease appears or is identified and/or a need for medication arises after inclusion but before initiation of the study.

Disease during conclusion of the study

Ages: 22 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Insulin stimulated muscle glucose uptake | Through study completion, approx. 1 year.
  Muscle glucose uptake during insulin stimulation in recovery from exercise (insulin sensitivity) will be determined based on Fick's principle. Thus, femoral arterio-venous difference (av difference) in blood glucose concentration will be multiplied by femoral arterial leg blood flow.

SECONDARY OUTCOMES:
Insulin stimulated muscle protein synthesis | 1-2 year.
  Muscle protein synthesis during insulin stimulation in recovery from exercise will be determined based on incorporation of 13C6-phenylalanine in muscle biopsies. Unit of measure is fractional synthesis rate (FSR) in percentage per hour (%/h).
Posttranslational modification of proteins in muscle biopsies | 5 years
  The obtained muscle samples will be subjected to mass spectrometry-based phosphoproteomic analysis. This measurement shows posttranslational modification that regulates protein function and will reveal the signalling network underlying the interventions studied. Unit of measure is log2-transformed arbitrary units.

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen FP Wojtaszewski, Professor, Principal Investigator — Department of Nutrition, Exercise and Sports, Faculty of Science, University of Copenhagen, Denmark
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No